CLINICAL TRIAL: NCT07013045
Title: Comparison of the Effects of Structured Neuromuscular Exercise Training and Neuromuscular Exergaming Program in Adolescents Diagnosed With Familial Mediterranean Fever
Brief Title: Comparing Structured Neuromuscular Exercise and Exergaming Program in Adolescents With Familial Mediterranean Fever
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Asya Albayrak, MSc, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fmfthesis
Record Dates: First submitted 2025-05-08; First posted 2025-06-10 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-05

CONDITIONS: Familial Mediterranean Fever (FMF )
Keywords: Familial Mediterranean Fever; Neuromuscular exercise; exergame
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Neuromuscular Exercise Training Group (Experimental): In the Structured Neuromuscular Exercise group, the exercise program will be implemented under the supervision of a physiotherapist for 12 weeks, twice a week, in patients diagnosed with FMF.
  Interventions: Other: Structured Neuromuscular Exercise Group
- Neuromuscular Exergaming Program Group (Experimental): In the Neuromuscular Exergaming program, the same exercises included in the Structured Neuromuscular Exercise group will be applied to patients diagnosed with FMF through an exergaming format, under the supervision of a physiotherapist, for 12 weeks, twice a week.
  Interventions: Other: Neuromuscular Exergaming Program Group

INTERVENTIONS:
Other: Structured Neuromuscular Exercise Group — In the Structured Neuromuscular Exercise group, the exercise program will be administered to patients diagnosed with FMF twice a week for 12 weeks under the supervision of a physiotherapist. The exercises will be performed using a balance board and will include sitting, standing, lunge, modified push-up, and plank positions.
  Arms: Structured Neuromuscular Exercise Training Group
Other: Neuromuscular Exergaming Program Group — In the Neuromuscular Exergaming group, patients diagnosed with FMF will perform the same exercises as those in the structured neuromuscular exercise program, delivered in an exergaming format using the Smart Exercise Board (SEG-Board). The program will be conducted under the supervision of a physiotherapist, twice weekly for 12 weeks, and will include exercises performed in sitting, standing, lunge, modified push-up, and plank positions.
  Arms: Neuromuscular Exergaming Program Group

SUMMARY:
Familial Mediterranean Fever (FMF) is an autosomal recessive, autoinflammatory disease characterized by recurrent fever attacks and inflammation of the serous membranes. FMF is defined by short, self-limiting inflammatory attacks that typically resolve within 1-3 days, and classic symptoms during an attack include fever, abdominal pain, chest pain, joint pain, and swelling.

Adolescents with chronic illnesses face numerous challenges in participating in physical activity, and often the disease itself leads to deconditioning and a decline in functional ability. Previous studies have reported that adolescents with FMF have lower cardiorespiratory fitness, exercise capacity, and muscle strength compared to their healthy peers. Even during attack-free periods, children experience high levels of fatigue, lower motivation and activity levels, and problems with concentration.

In the literature, there is evidence that physical activity and exercise programs are safe and feasible in rheumatic diseases such as Juvenile Systemic Lupus Erythematosus, Juvenile Idiopathic Arthritis, Juvenile Fibromyalgia, and Juvenile Dermatomyositis. These programs have been shown to improve patients' functional capacities, physical fitness, and reduce fatigue. However, only one study has been found regarding the effectiveness of physical activity and exercise programs in patients with FMF. This study compared the effectiveness of physical activity counseling and a 12-week online aerobic dance program conducted twice a week. It was found that both interventions led to positive improvements in functional capacity and physical fitness in children and adolescents with FMF, and aerobic dance was found to be feasible in this population. Accordingly, it is evident that further studies comparing the effects of different types of exercise in adolescents with FMF are needed in the literature.

Neuromuscular exercise is defined as a type of training that aims to improve the ability to generate controlled movement through coordinated muscle activation by enhancing various parameters such as muscle strength, flexibility, balance, and agility. Neuromuscular training programs conducted over 6-12 weeks have been shown to positively affect performance-related parameters in adolescent athletes from different sports disciplines, improve motor skills and motor control, enhance balance, proprioception, and core stabilization, reduce injury incidence, and improve both health- and skill-related physical fitness parameters.

Exergaming, derived from the combination of exercise training and video gaming, has gained significant popularity over the past few decades. In the literature, it has been found to improve muscular fitness and physical activity in obese children and adolescents, reduce the perception of fatigue and dyspnea in patients with Cystic Fibrosis, and be a safe option in various conditions with impaired neuromotor control, such as Down Syndrome, Developmental Coordination Disorder, and Cerebral Palsy. However, no study has been found investigating the effectiveness of exergaming in adolescents with FMF.

The aim of our study is to compare the effects of structured neuromuscular exercise training and a neuromuscular exergaming program in adolescents diagnosed with FMF.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 12 and 18 years
* Diagnosed with FMF at least 6 months ago at the Istanbul Faculty of Medicine, Pediatric Rheumatology Clinic
* Receiving routine medical treatment for FMF
* Being in an attack-free period
* Being willing to participate in the study

Exclusion Criteria:

* Having any chronic systemic disease other than FMF
* Having balance problems of vestibular or neurological origin
* Positive Fukuda (Unterberger) Test
* Having visual or hearing impairments
* Presence of scoliosis, leg length discrepancy, or recent lower extremity surgery
* Development of amyloidosis
* Presence of acute pain due to any cause

Withdrawal Criteria:

* Lack of cooperation with the exercise program
* Missing three consecutive exercise sessions

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
10-Stair Climb Test (10-SCT) | From enrollment to the end of treatment at 12 weeks
  The 10-SCT is commonly used to assess functional capacity in adolescents with chronic rheumatic diseases. During the test, participants will be asked to climb 10 steps (14x28x120 cm) as quickly as possible. The time taken to ascend the stairs will be recorded in seconds using a stopwatch.
6-Minute Walk Test (6MWT) | From enrollment to the end of treatment at 12 weeks
  The 6MWT is a simple, easy-to-administer, and well-tolerated test that reflects the submaximal level of functional capacity. It measures the distance a patient can walk quickly on a hard, flat surface within six minutes. Participants will be instructed on how to perform the test, and the distance walked in six minutes will be recorded in meters. The 6MWT will be used to assess the functional capacity of the participants.
30 Second Sit-to-Stand Test | From enrollment to the end of treatment at 12 weeks
  The 30SST is one of the tests used to assess lower extremity functional strength and performance in adolescents. During the test, participants will sit in the center of an armless chair with a seat height of 45 cm, feet flat on the floor, and arms crossed over their chest. Upon the evaluator's command, they will be instructed to stand up fully and sit back down using both lower limbs, completing as many sit-to-stand-to-sit cycles as possible within 30 seconds. Participants will also be instructed to perform at their maximum effort. The 30SST will be used to evaluate the functional performance of the lower extremities.

SECONDARY OUTCOMES:
FitnessGram Physical Activity Test Battery- Curl-up Test | From enrollment to the end of treatment at 12 weeks
  The curl-up test will be used to assess the abdominal muscle strength and endurance of the participants. The test will begin with the patient lying supine on an exercise mat, knees flexed at approximately 140°, feet flat on the floor, and legs slightly apart. Arms will be positioned parallel to the body and the floor, with palms placed flat on the ground and fingers extended. The goal of the test is to perform as many curl-ups as possible at a controlled pace. The rhythm of the test will be set to 20 curl-ups per minute, or one curl-up every 3 seconds. A maximum of 75 curl-ups will be counted. The test will end when the participant completes 75 curl-ups, fails to perform two consecutive repetitions correctly, or is unable to continue.
FitnessGram Physical Activity Test Battery- Push-up Test | From enrollment to the end of treatment at 12 weeks
  The push-up test will be used to assess upper extremity muscle strength and endurance. The test will begin with the patient in a prone position on an exercise mat, with hands placed at or slightly wider than shoulder-width apart, fingers extended, palms flat on the floor, and legs slightly apart. During the test, participants will lower their torso toward the floor by bending their elbows to approximately 90°, then push themselves back up to the starting position. The pace will be set at 20 push-ups per minute, or one push-up every 3 seconds. The test will be terminated if the participant makes two errors.
FitnessGram Physical Activity Test Battery- Trunk Lift Test | From enrollment to the end of treatment at 12 weeks
  The trunk lift test will be used to assess trunk extensor muscle strength and flexibility. The test will begin with the patient lying in a prone position on an exercise mat, with hands placed under the thighs. During the test, participants will slowly and in a controlled manner lift their upper body up to a maximum height of 12 inches (30.48 cm). At the end of the test, the distance between the participant's chin and the floor will be measured with a tape measure and recorded in centimeters.
FitnessGram Physical Activity Test Battery- Back-Saver Sit and Reach Test | From enrollment to the end of treatment at 12 weeks
  This test allows for the assessment of each leg separately, enabling the identification of any asymmetry in hamstring flexibility and helping to prevent knee hyperextension. The back-saver sit and reach test will be used to assess hamstring flexibility in patients. A test box is required for the procedure, measuring 35 cm in length, 45 cm in width, and 32 cm in height, with a top plate measuring 50 cm in length and 45 cm in width placed on top. During the test, participants will remove their shoes and sit in front of the test box. One leg will remain extended while the other is flexed. Participants will place one hand on top of the other and reach forward four times, holding the fourth reach for one second. The procedure will be repeated for the opposite leg. The distance reached will be recorded in centimeters.
Progressive Aerobic Cardiovascular Endurance Run (PACER) | From enrollment to the end of treatment at 12 weeks
  The PACER test is a modified version of the 20-meter shuttle run test and consists of multiple stages. It will be used to assess the aerobic capacity of the participants. During the test, patients will be asked to run back and forth between two cones placed 20 meters apart, following a pre-recorded audio cue set to music standardized by the Cooper Institute. The test begins at a slow pace and progressively increases in speed each minute. The test will be terminated when the participant can no longer maintain the required pace for their current level. If a participant fails to reach the cone at the sound of the beep for the first time, they will be instructed to continue running in the opposite direction and try to maintain the rhythm. At the end of the test, the total number of laps completed, including the lap that could not be completed, will be recorded.
Kinvent K-Plate Measurement System | From enrollment to the end of treatment at 12 weeks
  The KPlate, included in the Kinvent Measurement Set, will be used to evaluate the patients' static and dynamic balance.
Digitsole Pro® System | From enrollment to the end of treatment at 12 weeks
  The Digitsole Pro® system is capable of measuring walking patterns and gait variables under real-life conditions. The smart insoles of Digitsole Pro® can be placed inside any shoe, allowing for the measurement of spatial, temporal, and kinematic gait parameters. Gait profile of the patients will be assessed using Digitsole Pro®.
Fatigue Assessment Scale | From enrollment to the end of treatment at 12 weeks
  The Fatigue Assessment Scale is a 10-item questionnaire that includes five questions on physical fatigue and five on mental fatigue. It will be used to evaluate the fatigue levels of the patients.
Kinvent K-Pull Measurement System | From enrollment to the end of treatment at 12 weeks
  The K-Pull device, included in the Kinvent Measurement Set, will be used to assess the quadriceps and hamstring muscle strength of the patients.
Physical Activity | From enrollment to the end of treatment at 12 weeks
  The physical activity levels of the patients will be monitored using a smartwatch. The participants' step counts will be recorded via a smartwatch for a period of 3 months.
Exercise Satisfaction | From enrollment to the end of treatment at 12 weeks
  Patients' satisfaction levels will be assessed with Numerical Rating Scale. A score of 0 indicates no satisfaction from exercise, while a score of 10 indicates very high satisfaciton from exercise.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No